CLINICAL TRIAL: NCT00561912
Title: Phase II Study of Low Dose Decitabine (5-Aza-Deoxycytidine) With Interferon Alfa-2b in Advanced Renal Cell Carcinoma
Brief Title: Low Dose Decitabine + Interferon Alfa-2b in Advanced Renal Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0962
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Results first posted 2011-12-26 (Estimated); Last update posted 2011-12-26 (Estimated); Status verified 2011-11

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal Cell Carcinoma; Renal Cell Cancer; Clear Cell; Kidney; Decitabine; Dacogen; 5-Aza-Deoxycytidine; Interferon Alfa-2b; Intron A®; RCC
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Decitabine; Interferon alpha-2; Introns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Decitabine + Interferon Alfa-2b (Experimental): Decitabine 15 mg/m^2 intravenous (IV) daily over one hour for 5 days + Interferon Alfa-2b 0.5 million Units Subcutaneously Twice Daily Continuously, as of Cycle 3, Day 1.
  Interventions: Drug: Decitabine; Drug: Interferon Alfa-2b

INTERVENTIONS:
Drug: Decitabine — 15 mg/m^2 IV Daily over one hour for 5 days
  Other Names: 5-Aza-Deoxycytidine; Dacogen
Drug: Interferon Alfa-2b — 0.5 million Units Subcutaneously Twice Daily Continuously. Interferon Alfa-2b will be added on cycle three, day one.
  Other Names: Intron A®

SUMMARY:
Primary Objective:

* To determine the progression-free survival (PFS) times for patients with advanced renal cell carcinoma (RCC) treated with decitabine and interferon alfa-2b.

Secondary Objectives:

* To determine the toxicity of the combination of decitabine and interferon alfa-2b at the proposed dose and schedule in patients with advanced RCC
* To determine overall response by Response Evaluation Criteria in Solid Tumors (RECIST) criteria for patients with advanced RCC treated with decitabine and interferon alfa-2b.
* To determine the overall survival times for patients with advanced RCC treated with decitabine and interferon.
* To study the effects of decitabine and interferon alfa-2b on DNA methylation and gene expression in patients' tumor and non-tumor tissues and their correlation with clinical outcomes.
* To characterize the modulation of cellular immunity induced by the combination of decitabine and interferon alfa-2b in patients with advanced RCC and to correlate these results with clinical outcomes.

DETAILED DESCRIPTION:
THE STUDY DRUGS:

Decitabine is designed to slow tumor growth and may cause death of cancer cells.

Interferon alfa-2B is designed to activate your immune system, which may help keep tumors from growing, and may shrink tumors.

STUDY TREATMENT:

If you are found to be eligible to take part in this study, you will receive decitabine by vein over 1 hour on Days 1-5 of each cycle. A cycle in this study is 28 days long. All treatments with decitabine will take place at M. D. Anderson.

Once you have completed 2 cycles of decitabine (on Day 1 of Cycle 3), you will begin taking interferon alfa-2b twice each day (morning and afternoon) while continuing the same 5-day dosing schedule for decitabine. Interferon alfa-2b will be given as a subcutaneous (just under the skin) injection. It can be given by yourself or a caregiver at home or by your local doctor. You and your caregiver will be taught how to do the injection.

STUDY VISITS:

You will have the following tests/procedures performed during clinic visits.

On Day 1 of each cycle:

* You will have a physical exam, including measurement of your vital signs and weight.
* You will be asked about any medications or treatments you may be currently receiving.
* You will have a performance status evaluation.
* You will be asked about any side effects you may have experienced since your last visit. You will have blood drawn (about 1 teaspoon) for routine testing.

Beginning in Cycle 3, you will be required to return to the clinic around Day 14 of each cycle to have the following tests:

* You will have blood drawn (about 1 teaspoon each time) once a week for routine tests. If you do not experience severe side effects during Cycles 3 and 4, you will no longer be required to have weekly routine blood testing. Instead, you will return to have routine blood drawn on Day 1 of each cycle. This once-weekly schedule will restart if you experience severe side effects in Cycle 5.
* You will have a CT or MRI scan to check the status of the disease.
* Your vital signs will be measured
* You will be asked about any side effects you may have experienced since your last visit.

LENGTH OF STUDY:

You will continue taking the study drug combination unless the disease gets worse, you develop an illness that does not allow you to continue receiving the study therapy, or you experience any intolerable side effects. If any of these things occur, you will be removed from this study.

This is an investigational study. Decitabine is FDA approved and commercially available for the treatment of myelodysplastic syndrome (MDS). Interferon alfa-2b is FDA approved and commercially available for the treatment of several types of cancer, such as malignant melanoma, hairy cell leukemia, and non-Hodgkin's lymphoma. Their use together in this study in the treatment of PRC is investigational and authorized for use in research only.

Up to 60 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed clear cell renal carcinoma that is metastatic or unresectable. In the absence of metastatic disease, patients who are deemed unresectable or inoperable will have a documented surgical opinion confirming this. Surgical opinion will be rendered either by surgical consultation or after presentation at our interdisciplinary conference. Patients with locally recurrent RCC are eligible, if surgical resection of local recurrence is not feasible or is refused by patient.
* Patients with locally advanced unresectable RCC should have measurable or evaluable metastatic disease to be eligible for the protocol. Patients with bilateral renal cancer are eligible as long as both cancers are of clear cell type and patients have metastatic or unresectable disease.
* Patients may have received up to two prior anti-cancer therapies (including receptor tyrosine kinase inhibitors or cytokine therapy) but no prior chemotherapy for renal cell carcinoma. Patients should have received prior standard therapy, or otherwise deemed ineligible for such therapies.
* Patients must have measurable or clinically evaluable disease as defined by RECIST criteria.
* Patients must be >/= 14 days beyond the last administration of anti-cancer therapy, and must have recovered from the toxicities of prior therapy.
* Patients must be >/= 18 years of age.
* ECOG performance status </= 2 (Karnofsky >/= 60%).
* Patients must have adequate organ and marrow function, measured within 14 days of study entry, as defined below:

  * All Patients: Absolute neutrophil count >/= 1,500/microL; Platelets >/= 100,000/microL; Creatinine (serum) </= 2.0 mg/dL
  * Patients without liver metastases: Total bilirubin </= 1.5 mg/dL; AST(SGOT)/ALT(SGPT) </= 2.5 X Institutional Upper Limit of Normal (IULN)
  * Patients with liver metastases: Total bilirubin </= 1.5 x IULN; AST(SGOT)/ALT(SGPT) </= 5 x IULN
* The effects of decitabine and interferon on the developing human fetus are unknown. For this reason and because chemotherapy agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Female patients of childbearing potential should have a normal plasma beta human chorionic gonadotropin (betaHCG).
* Patients must give written informed consent prior to initiation of therapy in keeping with the policies of the institution. Patients with a history of major psychiatric illness must be judged able to fully understand the investigational nature of this study and the risks associated with the therapy.

Exclusion Criteria:

* Patients with active autoimmune disorders or who are receiving immunosuppressive therapy (including steroids or methotrexate) for any indication.
* Patients may not receive any other investigational agents within two weeks of study entry. Patients may not receive any other investigational agents while on study.
* Patients who have had major surgery within 2 weeks prior to entering the study, or have otherwise not adequately recovered from prior surgery.
* Patients who have had palliative radiation therapy within 1 week prior to entering the study.
* Patients with untreated or symptomatic brain metastases.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or potentially life-threatening cardiac arrhythmia.
* Psychiatric illness or social situations which in the opinion of the investigator could interfere with the completion of the proposed treatment.
* Pregnant women are excluded from this study because decitabine is an antimetabolite with the potential for teratogenic or abortifacient effects and interferon alfa-2b has abortifacient activity in animal studies. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with decitabine, breastfeeding should be discontinued if the mother is treated with decitabine or decitabine and interferon.
* Because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, patients known to be HIV-positive and receiving anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with the study agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana M. Aparicio, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 2 patients registered to the trial between the dates 31 October 2007 and 29 July 2008.
Pre-assignment Details: The trial was terminated early due to slow accrual and unavailable treatment agent.
Period: Overall Study
Arm/Group | Decitabine + Interferon Alfa-2b
Started | 2
Completed | 1
Not Completed | 1
Not completed — ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Decitabine + Interferon Alfa-2b
Number analyzed (Participants) | 2
Age Continuous [Mean (Full Range); unit: years] | 53 [47 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Times
Description: Progression-free survival (PFS) times for participants with advanced renal cell carcinoma (RCC) treated with decitabine and interferon alfa-2b where PFS is defined as starting from day one of the treatment combination to disease progression or death for any reason, measured in weeks.
Time Frame: From treatment start or until disease progression or death for any reason, at least 16 weeks
Population: With one of the two participants ruled ineligible and inevaluable, there was insufficient data for statistical evaluation.
Measure: Number; unit: Weeks
Arm/Group | Decitabine + Interferon Alfa-2b
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Decitabine + Interferon Alfa-2b
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No